CLINICAL TRIAL: NCT06186648
Title: A Phase 2 Study Evaluating the Bispecific CD3xCD20 Antibody GLOfitamab in Combination With Rituximab or Obinutuzumab Plus Cyclophosphamide, Doxorubicin, Vincristine and Prednisone (CHOP) in Patients With RIchter Syndrome as Frontline therapY. A FILO Study
Brief Title: Evaluation of Treatment by Glofitamab in Combination With Rituximab or Obinutuzumab Plus CHOP in Patients With RIchter Syndrome
Acronym: GLORIFY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FILOCLL015 - GLORIFY
Record Dates: First submitted 2023-12-06; First posted 2024-01-02 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Richter Syndrome
MeSH Terms: interventions — glofitamab; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glofitamab + Obinutuzumab (Experimental): cf Intervention
  Interventions: Drug: Glofitamab + Obinutuzumab

INTERVENTIONS:
Drug: Glofitamab + Obinutuzumab — Duration of each cycle is 21 days. Cycle 1: R-CHOP Cycle 2: G-CHOP + glofitamab (at this cycle onnly, Obinutuzumab will be injected instead of Rituximab in order to decreased the risk of cytokine released syndrome) Cycle 3-6: R-CHOP + glofitamab Cycle 7-8: glofitamab alone

SUMMARY:
This is a national clinical trial, multicentric (28 centers), non-randomized phase 2 study.

Population: Patients with previously untreated Richter's syndrome (RS), defined as the occurrence of an aggressive lymphoma (of diffuse large B-cell lymphoma histology) in a patient with chronic lymphocytic leukemia (CLL).

Study treatment:

The duration of each cycle is 21 days.

Cycle 1:

Participants will receive standard of care doses of R-CHOP in cycle 1 as follows:

* Rituximab 375 mg/m² IV Day 1
* Cyclophosphamide 750 mg/m² IV Day 1
* Doxorubicin 50 mg/m² IV Day 1
* Vincristine 1.4 mg/m² [capped at 2.0 mg] IV Day 1
* Prednisone 60 mg/m2 per day PO Day 1-5

Cycle 2:

In order to minimize cytokine release syndrome (CRS), participants will then receive G-CHOP as cycle 2 (with obinutuzumab) and glofitamab:

* Obinutuzumab 1000 mg single dose IV Day 1
* Cyclophosphamide 750 mg/m² IV Day 1
* Doxorubicin 50 mg/m² IV Day 1
* Vincristine 1.4 mg/m² [capped at 2.0 mg] IV Day 1
* Prednisone 60 mg/m2 per day PO Day 1-5
* Glofitamab : administered intravenously (IV) as a step-up dose on Days 8 (2.5 mg) and 15 (10 mg)

Cycle 3-6:

Participants will receive standard of care doses of R-CHOP and Glofitamab as follows:

* Rituximab 375 mg/m² IV Day 1
* Cyclophosphamide 750 mg/m² IV Day 1
* Doxorubicin 50 mg/m² IV Day 1
* Vincristine 1.4 mg/m² [capped at 2.0 mg] IV Day 1
* Prednisone 60 mg/m2 per day PO Day 1-5
* Glofitamab : 30 mg IV Day 8

Cycle 7 and 8 (only for patient in Complete Response or Partial response after Cycle 6):

Cycle 7 and 8 consist of 2 infusions of glofitamab only at D8C7 and D8C8:

● Glofitamab : 30 mg IV Day 8

Primary endpoint Percentage of participants with a complete response as assessed by the investigator using the Cheson IWG 2014 Lugano Classification (i.e. Deauville scale 1-3) after 6 cycles of R/G-CHOP + glofitamab or at permanent treatment discontinuation.

End of treatment is defined as after 6 cycles of R/G-CHOP + glofitamab. Permanent treatment discontinuation is defined as the discontinuation of all treatments (R/G-CHOP, glofitamab).

DETAILED DESCRIPTION:
Study design :

Open label, multicenter phase 2 trial

Population:

Patients with previously untreated Richter's syndrome (RS), defined as the occurrence of an aggressive lymphoma (of diffuse large B-cell lymphoma histology) in a patient with chronic lymphocytic leukemia (CLL).

Primary objective:

The primary objective is to determine the objective response regarding the RS to 6 cycles of R/G-CHOP + glofitamab in patients with RS.

Secondary objectives:

The secondary objectives are to investigate the safety and toxicity of 6 cycles R/G-CHOP + glofitamab, the response to 6 cycles of R/G-CHOP + glofitamab and the patient outcome.

Sample size : 40 patients Length of study: Inclusion period: 18 months Treatment duration: 6 months (24 weeks) Follow-up period: 12 months Duration of the study: 36 months

Study treatment:

The duration of each cycle is 21 days.

Cycle 1:

Participants will receive standard of care doses of R-CHOP in cycle 1 as follows:

Rituximab 375 mg/m² IV Day 1 Cyclophosphamide 750 mg/m² IV Day 1 Doxorubicin 50 mg/m² IV Day 1 Vincristine 1.4 mg/m² [capped at 2.0 mg] IV Day 1 Prednisone 60 mg/m2 per day PO Day 1-5

Cycle 2:

In order to minimize cytokine release syndrome (CRS), participants will then receive G-CHOP as cycle 2 (with obinutuzumab) and glofitamab:

Obinutuzumab 1000 mg single dose IV Day 1 Cyclophosphamide 750 mg/m² IV Day 1 Doxorubicin 50 mg/m² IV Day 1 Vincristine 1.4 mg/m² [capped at 2.0 mg] IV Day 1 Prednisone 60 mg/m2 per day PO Day 1-5 Glofitamab : administered intravenously (IV) as a step-up dose on Days 8 (2.5 mg) and 15 (10 mg)

Cycle 3-6:

Participants will receive standard of care doses of R-CHOP and Glofitamab as follows:

Rituximab 375 mg/m² IV Day 1 Cyclophosphamide 750 mg/m² IV Day 1 Doxorubicin 50 mg/m² IV Day 1 Vincristine 1.4 mg/m² [capped at 2.0 mg] IV Day 1 Prednisone 60 mg/m2 per day PO Day 1-5 Glofitamab : 30 mg IV Day 8 Evaluation will be performed after C4 and C6 (see 6.2.3. and 6.2.4.). Responding patients with response (CR or PR according to Cheson IWG 2014 Lugano Classification (i.e. Deauville scale 1-3)) after C6 will receive two more infusions of glofitamab (day 8 of C7 and C8).

Cycle 7 and 8:

Cycle 7 and 8 consist of 2 infusions of glofitamab only at D8C7 and D8C8:

Glofitamab : 30 mg IV Day 8

Study procedures:

Screening period :

Assessments may be done up to 28 days before the treatment start and will include:

Clinical assessments Medical history including demographics, previous and current diseases, medications included previous CLL treatment(s) Physical examination (B symptoms, weight, height), tumor lesion assessment including peripheral nodes location and two dimensional diameters, vital signs (pulse, blood pressure, body temperature) Binet staging (appendix 3) ECOG performance status (appendix 4) Ann Arbor staging (appendix 5) Assessment of the international Prognostic Index (IPI) (appendix 6) Determination of the CIRS score (appendix 7) Standard laboratory assessments Hematology Biochemistry Other exams HIV 1-2, HBV and HCV serology (Ag HBs, Ac anti-HBs, Ac anti-HBc, Ac anti-VHC), SARS-COV-2 serology and PCR Pregnancy test (beta-HCG) for women of child-bearing potential Coagulation test (fibrinogen, APTT, PT) Specific assessments Immunophenotyping (including CD38) of peripheral lymphocytes and Matutes RMH score Karyotype and 4-color FISH analysis for: 17p13 deletion, 11q22 deletion, 13q14 deletion and trisomy 12 of either blood or marrow CLL cells IGHV mutational status on CLL samples (at baseline or before). IGHV status should also be performed on the Richter specimen DNA in order to determine the clonal relationship between RS and CLL.

TP53 gene sequencing according to ERIC recommendation (on CLL cells). Bone marrow biopsy Imaging exams Whole-body CT scan (thorax, abdomen, pelvis) and measurement in two perpendicular dimensions and response assessments according to the revised Lugano criteria (appendix 1) Whole body PET-scan with SUV measurement and response assessments according to the revised Lugano criteria (appendix 1).

Other exams 12-lead ECG Assessment of left ventricular ejection function by either cardiac ultrasound or isotopic ventriculography

Treatment period :

Before each cycle (R/G-CHOP)

Clinical assessment:

Physical examination Concomitant medications Adverse events, serious adverse events and adverse events of special interest Hematology Biochemistry Before each cycle (Glofitamab alone)

Clinical assessment:

Vital signs (pulse, blood pressure, body temperature) Concomitant medications Adverse events, serious adverse events and adverse events of special interest Hematology Biochemistry Electrolytes (sodium, potassium, calcium, phosphore) Total protein, glycemia, urea, uric acid, serum creatinine and creatinine clearance (Cockroft and Gault formula) Bilirubin, ASAT, ALAT, GGT, alkaline phosphatases LDH C-reactive protein After 4 cycles of R/G-CHOP + glofitamab (W12) and after 6 cycles of R/G-CHOP + glofitamab (W18)

Clinical assessment:

Physical examination (B symptoms, weight, height, ECOG performance status), tumor lesion assessment including peripheral nodes location and two dimensional diameters Vital signs (pulse, blood pressure, body temperature) Writing test (C6 only) Concomitant medications Adverse events, serious adverse events and adverse events of special interest Hematology Biochemistry

Imaging exams Whole-Body CT scan Whole body PET-scan with suv measurement and response assessment according to the revised Lugano criteria (appendix 1) will also be performed.

Only after 6 cycles of R/G-CHOP + glofitamab (W18) Bone marrow biopsy only if CR criteria obtained in both CT scan and PET. Follow up assessments The follow-up will be performed every 3 months for 12 months (FU3, FU6, FU9, FU12) after the end of last treatment by glofitamab (C8D8) or if patient stopped treatment prematurely without initiate a new treatment.

End of treatment (EOT):

A visit will be performed within 30 days after the last administration of study treatment for patient stop treatment prematurely and Withdrawn of the study A discontinuation/withdrawal form will be sent to the Filo secretary and head of project.

For patient continue follow up visits no EOT is required.

End of study (EOS):

The end of study becomes effective after the end of last study visit of last patient enrolled and performed the FU12 visit.

The end of study visit corresponds to the last follow-up visit (FU12). For patient withdraw during follow up period, no end of study visit is required.

Observational study:

For all patient without withdrawn at FU12 visit (see paragraph 9.2 definition of withdrawal):

After this last study visit and if patient consents, the Survival date will be collected every year in the eCRF (Survival date and/or event date form) until death, for analyse the survival:

Date of last news. Patient status: alive/death/lost of sight Patient response. Initiation of new treatment.

Investigational product:

Obinutuzumab (Gazyvaro®) Obinutuzumab is a humanized glycoengineered type II anti-CD20 monoclonal antibody that recognizes the CD20 antigen present on normal and malignant B cells and is being developed for the treatment of hematological malignancies including NHL and CLL.

Glofitamab:

Glofitamab is a "2:1" T-cell bispecific humanized monoclonal antibody that binds to human CD20 on B cells through two fragment antigen-binding domains, and to the human CD3 epsilon subunit (CD3e) of the T-receptor (TCR) complex on T cells through a single Fab domain.

Safety :

Patient safety will be assessed based on clinical and laboratory evaluations, physical examinations, vital signs, and monitoring of adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of chronic lymphocytic leukemia or small lymphocytic lymphoma according to the revised iwCLL criteria with biopsy proven transformation to CD20 positive diffuse large B-cell lymphoma, consistent with RS according to the 2016 WHO classification
2. A fresh or archival tissue biopsy is mandatory
3. Previous therapy for CLL is allowed (but no prior therapy for RS)
4. Age greater than or equal to 18 years and less or equal to 80 years
5. ECOG performance status 0-2
6. Participants must have at least one measurable target lesion (≥ 1.5 cm) in its largest dimension by computed tomography (CT) scan. Measurable disease, defined as at least one bi-dimensionally measurable nodal or tumor lesion, defined as > 1.5 cm in its longest dimension or PET-CT with at least one hypermetabolic lesion. Patients without measurable disease but with proven bone marrow infiltration by the RS are eligible.
7. Patients must meet the following hematologic criteria at screening, unless they have significant bone marrow involvement of either CLL or RS cells confirmed on biopsy: absolute neutrophil count ≥ 1.5 G/L, hemoglobin >10 g/dL, and platelet count ≥75 G/L independent of transfusion within 7 days of screening
8. Subject must have adequate coagulation tests: Prothrombin Time > 50%, Fibrinogen > 1 g/L
9. Adequate liver function: Total bilirubin ≤ 1.5 x ULN; Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 x ULN
10. Adequate left ventricular ejection function (> 50 %)
11. Adequate renal function: creatinine clearance calculated by MDRD/Cockcroft-Gault formula of ≥ 40 mL/min
12. Negative serologic or PCR test results for acute or chronic HBV infection
13. Negative test results for HCV and HIV (Patients who are positive for HCV antibody must be negative for HCV by PCR to be eligible for study participation)
14. Prior vaccination to the SARS-Cov-2 virus and and SARS-CoV-2 PCR testing and negative result before study treatment administration at each treatment cycle
15. Negative serum or urinary pregnancy test within 7 days prior to study treatment in women of childbearing potential. Patients must agree to either remain completely abstinent or to use two effective contraceptive methods* until:

    * If the patient is a male: at least 3 months after pre-treatment with obinutuzumab or RCHOP or 2 months after the last dose of glofitamab, whichever is longer. Men must refrain from donating sperm during this same period
    * If patient is a female of childbearing potential: until at least 18 months after pre-treatment with obinutuzumab or RCHOP or 2 months after the last dose of glofitamab, whichever is longer
16. Ability to understand and the willingness to sign a written informed consent document. Patient must be willing and able to comply with protocol-mandated hospitalization upon administration of the first dose of glofitamab. Patient must also be willing to comply with all study-related procedures
17. Signed written informed consent
18. Patient covered by any social security system

Exclusion Criteria:

1. Patients with the Hodgkin variant of RS
2. Patients with previously treated for RS
3. Current or past history or presence of clinically relevant disorder affecting the central nervous system (CNS)
4. Ineligible to CHOP full dose for any reason
5. Previous treatment with a bispecific antibody
6. Current or past history of DLBCL in the CNS (confirmed by CSF analysis)
7. Steroids treatment (> 1 mg/kg/d for one week) before inclusion
8. History of anaphylactic reactions to human, chimeric, or mouse monoclonal antibodies or to any components of the product.
9. Prior allogeneic HSCT
10. Patients with known acute infection or reactivation of a latent infection, whether bacterial, viral (including, but not limited to, EBV, cytomegalovirus (CMV), hepatitis B, hepatitis C, HIV and SARS-CoV-2), fungal, mycobacterial, or other pathogens (excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics (for IV antibiotics this pertains to completion of last course of antibiotic treatment) within 4 weeks prior to the first study treatment.
11. History of other malignancies, except: i) malignancy treated with curative intent and with no recurrence over the last 3 years ii) adequately treated non-melanoma skin cancer without evidence of disease iii) adequately treated carcinoma in situ without evidence of disease
12. Prior solid organ transplantation
13. History of treatment-emergent immune-related adverse events associated with prior immunotherapeutic agents, as follows:

    * Grade ≥ 3 adverse events with the exception of Grade 3 endocrinopathy managed with replacement therapy
    * Grade 1-2 adverse events that did not resolve to baseline after treatment discontinuation
14. Current uncontrolled autoimmune disease*
15. History of human immunodeficiency virus
16. Hepatitis B or C seropositivity (unless clearly due to vaccination)
17. Pregnant or breastfeeding women
18. Unwilling or unable to participate in all required study evaluations and procedures.
19. Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form and authorization to use protected health information (in accordance with national and local subject privacy regulations)
20. Persons deprived of their liberty by judicial or administrative decision, persons subject to a legal protection measure (guardianship, curatorship, legal protection), persons under psychiatric care
21. Fertile male patients who cannot or do not wish to use an effective method of contraception, during and for 12 months after the final treatment used for the purposes of the study.
22. Patients with history of macrophage activation syndrome (MAS) / hemophagocytic lymphohistiocytosis (HLH)
23. LVEF < 50% as determined by echocardiography or multiple uptake gated acquisition (MUGA) scan, significant or extensive cardiovascular disease such as New York HeartAssociation Class III or IV cardiac disease or Objective Assessment Class C or D,myocardial infarction within the last 3 months, unstable arrhythmias, or unstable angina.
24. Abnormal screening laboratory values as defined as following: a) ALT (SGOT) and/or ALT (SGPT) and/or ALP ≥ 3 x upper limit of normal (ULN); b) Total bilirubin ≥ 1.5 x ULN, unless due to Gilbert's disease; c) Creatinine ≥ 2.0 x ULN or creatinine clearance < 40 mL/min (calculated).
25. Patient with history of confirmed progressive multifocal leukoencephalopathy (PML)
26. History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
27. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug
28. Major surgery or significant traumatic injury < 28 days prior to the obinutuzumab infusion (excluding biopsies) or anticipation of the need for major surgery during study treatment
29. Administration of a live, attenuated vaccine within 4 weeks before obinutuzumab infusion
30. Treatment with another investigational agent or participating in another trial within 30 days prior to entering the study
31. Clinically significant history of liver disease or cirrhosis
32. Pregnant or breast-feeding or intending to become pregnant during the study
33. No affiliation to social security
34. Inability to comply with protocol mandated hospitalization and restrictions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective response regarding Richter Syndrome to R/G-CHOP + glofitamab combination. | 6 cycles (each cycle is 21 days)
  Percentage of patients with a complete response (CR) assessed using the Cheson IWG 2014 Lugano Classification (i.e. Deauville scale 1-3)

SECONDARY OUTCOMES:
Safety and toxicity of the R/G-CHOP + glofitamab combination | Through treatment completion, an average of 8 months
  Advers events evaluation according to the Common Terminology Criteria for Adverse Events (CTCAE) v.5 and American Society for Transplantation and Cellular Therapy (ASTCT) Consensus grading for International Conference on Harmonization (ICANS) and Cytokine Release Syndrom (CRS)

CONTACTS AND LOCATIONS:
Overall Officials: Romain guièze, MD, Principal Investigator — Service d'hématologie clinique adulte et de thérapie cellulaire Etablissement : CHU Estaing
Locations (23):
- France (23):
  - Amiens-Picardie Chu, Amiens
  - Angers Chu, Angers
  - BAYONNE - CH de la Côte Basque - Hématologie, Bayonne
  - Clermont-Ferrand - Chu Estaing, Clermont-Ferrand
  - Grenoble - CHUGA - Hématologie Clinique, Grenoble
  - LILLE GHICL - Hôpital Saint Vincent de Paul, Lille
  - LILLE CHU - Hôpital Claude Huriez, Lille
  - LIMOGES - CHU Dupuytren 1, Limoges
  - LYON-Centre Léon Bérard, Lyon
  - MONTPELLIER - Hôpital Saint-Eloi - Hématologie Clinique, Montpellier
  - APHP - Hôpital Saint-Louis - Hématologie adultes, Paris
  - APHP - Hôpital Saint-Antoine - Hématologie et thérapie cellulaire, Paris
  - APHP - Hôpital Pitié Salpêtrière - Hématologie, Paris
  - Bordeaux Pessac, Pessac
  - LYON HCL - CH Lyon Sud, Pierre-Bénite
  - Reims Chu, Reims
  - RENNES - CHU Pontchaillou - Hématologie Clinique, Rennes
  - ROUEN - Centre Henri Becquerel - Service Hématologie Clinique, Rouen
  - Strasbourg - Icans, Strasbourg
  - Toulouse - IUCT Oncopole - Service d'Hématologie, Toulouse
  - TOURS - Hôpital Bretonneau, Tours
  - NANCY - CHU Brabois, Vandœuvre-lès-Nancy
  - VERSAILLES - Hôpital André Mignot, Versailles

IPD SHARING:
Plan to Share IPD: No